CLINICAL TRIAL: NCT05530733
Title: Clinical Effects of Pacifier Use in Preterm During Orogastric Tube Feeding: Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Yeliz Taşdelen, Principal investigator, Nurse, Research assistant, Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BEU-YTASDELEN-001
Record Dates: First submitted 2022-08-29; First posted 2022-09-07 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-03

CONDITIONS: Premature; Pacifiers; Tube Feeding; Neonatal Nursing
MeSH Terms: conditions — Premature Birth | interventions — Pacifiers; Milk, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pacifier only (Other): Participants in the pacifier-only group will get a pacifier five minutes prior to tube feeding. During feedings, a pacifier will be employed. Five minutes following the end of tube feeding, the pacifier application will be discontinued. The vital signs will be monitored prior to, during, and following feeding. Two hours after the feeding has finished, the volume of gastric residue will be controlled.
  Interventions: Procedure: Pacifier
- Pacifier with breast milk (Other): Five minutes prior to tube feeding, participants in the pacifier with breast milk group will get their own breast milk dripping pacifier. During feedings, a pacifier will be employed. Five minutes following the end of tube feeding, the pacifier application will be discontinued. The vital signs will be monitored prior to, during, and following feeding. Two hours after the feeding has finished, the amount of gastric residue will be controlled.
  Interventions: Procedure: Pacifier; Procedure: Breast milk
- standard care (no pacifier) (No Intervention): The premature babies in the standard care (no pacifier) will get standard care while being fed through an orogastric tube. The vital signs will be monitored prior to, during, and following feeding. Two hours after the feeding has finished, the amount of gastric residue will be controlled.

INTERVENTIONS:
Procedure: Pacifier — Pacifiers produced for premature babies will be used in the study. Pacifiers will be made of silicone material suitable for premature baby health and will not contain any harmful substances. A separate pacifier will be used for each baby, and pacifiers will be sterilized before use.
  Arms: Pacifier only; Pacifier with breast milk
Procedure: Breast milk — For babies assigned to the pacifier with breast milk group, their own breast milk will be applied by dripping 1 ml into the pacifier.
  Arms: Pacifier with breast milk

SUMMARY:
The purpose of the study was to assess how preterm babies' vital signs, feeding time, and gastric residual volume were affected by using a pacifier only or a pacifier with breast milk during orogastric tube feeding.

ELIGIBILITY:
Inclusion Criteria:

* Feeding with the orogastric tube
* Breastmilk along with formula (babies who receive more than 50% of their total feed in 24 hours from formula)
* Gestation week between 29+0 weeks and 34+0 weeks
* Weight of 1000 g or more

Exclusion Criteria:

* Receiving mechanical ventilator support
* Development of sepsis
* Presence of neurological disease
* Presence of chromosomal or congenital anomalies
* Presence of intraventricular bleeding
* Unstable physiological parameters
* No breast milk

Ages: 29 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Heart rate change | 5 minutes before tube feeding, during tube feeding and 5 minutes after tube feeding
  Heart rate will be measured 5 minutes before tube feeding, during tube feeding and 5 minutes after the end of tube feeding.
Respiratory rate change | 5 minutes before tube feeding, during tube feeding and 5 minutes after tube feeding
  Respiratory rate will be measured 5 minutes before tube feeding, during tube feeding and 5 minutes after the end of tube feeding.
Saturation level change | 5 minutes before tube feeding, during tube feeding and 5 minutes after tube feeding
  Saturation level will be measured 5 minutes before tube feeding, during tube feeding and 5 minutes after the end of tube feeding.
Feeding duration | measured with a stopwatch for 7 months.
  Each baby's tube feeding duration will be measured.
Gastric residual volume | Gastric residue will be measured 2 hours after the end of infant feeding.
  Gastric residue will be measured 2 hours after the end of infant feeding.

CONTACTS AND LOCATIONS:
Locations (1):
- Yeliz Taşdelen, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No